CLINICAL TRIAL: NCT00863356
Title: Trial of a Novel Chitosan Hemostatic Sealant in the Management of Complicated Epistaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HemCon Medical Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-I-Epistaxis-1
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Results first posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-09

CONDITIONS: Epistaxis
Keywords: Epistaxis; Chitosan; Hemostatic; Nose bleed; Nasal bleeding; Nasal pack; Sealant; ChitoFlex®; HemCon; HemCon® ChitoFlex Surgical Dressing; HemCon® Nasal Plugs; Biocompatible dressing
MeSH Terms: conditions — Epistaxis | interventions — Hemostatic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epistaxis Group (Experimental): Subjects presenting with epistaxis that have not been controlled by traditional nasal packing, or that recurred immediately upon removal of the nasal packing will be included in this study. Subject will be evaluated during the packing period to determine the effect of hemostasis. Chitosan coated packing will be removed after 48 hours. Subjects' nasal cavities will be examined endoscopically to evaluate bleeding control, morphological changes induced by the chitosan coated packing.
  One week after the removal of the packing, the patients will be endoscopically examined to assess the healing of the packed area, to monitor control of bleeding, and observe any potential delayed reaction to the packing material.
  Interventions: Device: 2009-I-Epistaxis-1

INTERVENTIONS:
Device: 2009-I-Epistaxis-1 — Trial of a Novel Chitosan Hemostatic Sealant in the Management of Complicated Epistaxis, 48 hour removal, 1 week follow-up.
  Other Names: Epistaxis; Chitosan; Chitin; Hemostatic; Nose bleed; Nasal bleeding; Nasal pack; Sealant; ChitoFlex®; HemCon; HemCon® ChitoFlex Surgical Dressing; HemCon® Nasal Plugs; biocompatible polysaccharide

SUMMARY:
Purpose:

This study is a prospective clinical trial to investigate the efficacy of a chitosan-coated nasal packing (ChitoFlex® used in conjunction with the HemCon Nasal Plug) in the management of difficult spontaneous epistaxis and to evaluate its healing effect on nasal mucosa.

The introduction of products that enhances hemostasis can have clinical advantages when associated with traditional nasal packing. These advantages include a better hemostatic control and the reduction of nasal packing duration. Furthermore, this study will help determine if there are any non-desirable effects that chitosan may have on the nasal cavity, such as the production of fibrosis and foreign body reaction.

DETAILED DESCRIPTION:
Epistaxis is a common reason for emergency department visits and otolaryngology referral. Management methods of epistaxis include nasal packing, chemical or electric cauterization, and arterial ligation or embolization.

There are numerous nasal packing products available in the market, and are used to stop or prevent nasal bleeding. The ideal nasal pack should be efficient in controlling bleeding, have antimicrobial properties and be well tolerated. Currently, there is no perfect nasal pack, but some are closer to ideal than others. Nasal packs can be classified into non-absorbable and absorbable nasal packs.

Recently, a new hemostatic product has been introduced in the market, and used as a military wound bandages, the ChitoFlex®. ChitoFlex® is made of chitosan, a naturally occurring, bio-compatible polysaccharide. Because chitosan has a positive charge, it attracts red blood cells, which have a negative charge. The red blood cells create a seal over the wound as they are drawn into the bandage, forming a very tight, coherent seal. The ChitoFlex® -dressing has been demonstrated by AATCC Test Method 100-2004, Evaluation of Antibacterial Finishes (Technical Manual of the America Association of Textile Chemists and Colorists) as an antibacterial barrier in laboratory testing with a variety of gram-positive and gram-negative bacterial organisms.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years.
* Epistaxis despite nasal packing or rebleeding after removal of the packing.

Exclusion Criteria:

* Patient unable or unwilling to provide informed consent.
* Prior diagnosis of disease or medical condition affecting the ability of blood to clot (e.g., hemophilia.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan H. Shikani, MD, FACS, Principal Investigator — Union Memorial Hospital
Locations (1):
- Union Memorial Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from a tertiary rhinology fellowship training clinic from January 2009 to November 2009.
Period: Overall Study
Arm/Group | Epistaxis Group
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Epistaxis Group
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 67 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: This Study Evaluates the Efficacy of HemCon Hemostatic Agent in Control of Complicated Epistaxis in Terms of % Success of Hemostasis. Success Will be Defined as Achieving Active Control of Bleeding Before Patient Leaves the Physicians Office.
Time Frame: Removal: 48 hours. Follow-up: 1 week.
Reporting Status: Not Posted

2. Secondary Outcome: This Study Evaluates the Benefits Acquired by the Use This New Product in Terms of Presence/Absence of Post-packing Tissue Scarring. This Will be Accessed by Endoscopic Examination of the Nasal Cavity Following Removal of HemCon Material.
Time Frame: Removal: 48 hours. Follow-up: 1 week.
Reporting Status: Not Posted

3. Primary Outcome: Hemostasis Success
Description: Successful hemostasis prior to leaving physician's office
Time Frame: From procedure to hemostasis.
Population: All enrolled subjects
Measure: Number; unit: percentage of participants
Arm/Group | Epistaxis Group
Number analyzed (Participants) | 20
percentage of participants | 20

ADVERSE EVENTS:
Arm/Group | Epistaxis Group
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No